CLINICAL TRIAL: NCT03063905
Title: The Effects of Opioid Taper on Opioid-Induced Hyperalgesia
Status: Terminated | Type: Observational
Why Stopped: funding expired
Sponsor: Georgetown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-0028; U01DA029580 (NIH)
Record Dates: First submitted 2017-02-08; First posted 2017-02-24 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Buprenorphine; Pain
Keywords: Opioid related disorders; Narcotic abuse
MeSH Terms: conditions — Pain; Opioid-Related Disorders; Narcotic-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opioid Taper: Patients tapering off their buprenorphine treatment
  Interventions: Drug: Buprenorphine
- Opioid Maintenance: Patients starting their buprenorphine treatment
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Patients taking buprenorphine to wean off an opiate addiction
  Other Names: Suboxone

SUMMARY:
Evidence to support the effectiveness of ongoing opioid therapy for the treatment of chronic non-malignant pain is lacking. In fact, data suggest that patient outcomes improve when tapered off opioid analgesics. To better understand the role opioid therapy plays in the experience of pain, we will study measured pain sensitivity in opioid dependent patients over the course of and 3 months following a standardized opioid taper. By isolating the effect of opioid taper in patients without pain, preliminary evidence of effect size can be used to guide clinicians treating patients with chronic pain.

DETAILED DESCRIPTION:
Chronic pain impacts the daily lives of fully one-third of Americans over the age of 45, with prevalence expected to increase as the population ages. In well-intended and industry-driven efforts to provide relief to chronic pain sufferers, the prescription of opioids has increased dramatically since the turn of the century, such that it is currently estimated that between 5 and 8 million Americans use opioids on a daily basis for chronic pain management. Yet, prescription opioid therapy for chronic pain is not an evidence-based intervention. In fact, as evaluation data accumulate, it is becoming clear that outcomes are often poorer for patients on opioid therapy, and that improvements are appreciated when tapered off the medications. In the midst of an "epidemic of prescription drug abuse" it is critical that opioid prescription practices be evidence-based and delivered "in the best possible manner that maximizes effectiveness and minimizes harm".

A theorized explanation for poorer outcomes (functionality, quality of life) for patients on opioid therapy is the phenomenon of opioid-induced hyperalgesia (OIH). Well-demonstrated in animal and inferred in patients, ongoing opioid use results in increased sensitivity to experimental pain, which, in the case of the chronic pain patient, is believed to interfere with (if not preclude) desired pain relief outcomes. However, the causal relationship between opioid discontinuation and OIH has received little empirical attention, such that it is not clear the degree to which opioid taper improves pain responses and outcomes, if at all. Evidence supporting that prescription opioids makes the pain experience worse for chronic pain patients would support a sea change in current practice of chronic opioid therapy.

Studying the direct effects of an opioid taper on pain responses in chronic pain patients is challenging; complicated by the reemergence of pain, variable compliance with taper and concomitant increased use of non-opioid pain medications, a controlled examination of pain responses during and following opioid detoxification is not immediately tenable in this patient population. Thus, funded is a proof-of concept trial to identify and characterize the direct effects of opioid detoxification on experimental pain responses in opioid-dependent patients without chronic pain to establish if, in fact, a notable effect size can be discerned. If supported, these findings will provide a foundation upon which to predict efficacy in patients with the more complicated picture of chronic pain.

Specifically, in a well-characterized sample of men and women seeking addiction treatment in a residential setting, experimental pain responses will be serially described over the course of and for three months following a standard observed opioid (buprenorphine) taper, and compared to those of matched control patients initiated on buprenorphine maintenance therapy. Pain responses will be measured with two valid and reliable experimental pain induction techniques commonly used to measure OIH (cold-pressor, quantitative sensory testing), and subject-level predictors of response identified.

ELIGIBILITY:
Inclusion Criteria:

1. between ages of 18-50
2. able to provide a positive urine toxicology test for heroin, morphine and/or methadone (and free of other drugs of abuse) upon treatment admission
3. without known background disease, including chronic or acute pain
4. otherwise in good physical and mental health, or in the care of a physician who is willing to take responsibility for such treatment
5. able to understand the purpose and instructions of the study, and provide informed consent as approved by the Western and Georgetown University Institutional Review Boards

Exclusion Criteria:

1. meet diagnostic criteria for an active substance use disorder other than opioids and nicotine
2. be acutely psychotic, severely depressed, and/or in need of inpatient psychiatric treatment
3. have a neurological (i.e. Raynaud's syndrome or symptomatic cold neuropathy) or psychiatric illness that would affect pain responses
4. have a history of heart disease, stroke, or a pacemaker or uncontrolled high blood pressure. Good cardiovascular health is stipulated to ensure subjects can tolerate the sympathetic nervous system responses associated with the pain induction procedures.
5. have sensory deficits at pain testing site resulting from medical conditions such as diabetes, alcoholic neuropathy, AIDS neuropathy, severe thyroid, and liver or kidney diseases

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Men and women seeking addiction treatment in a residential or outpatient setting
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Pain Threshold Response (in seconds) - Cold Pressor Test | 3 months
  To compare the effects of opioid taper with initiating buprenorphine maintenance therapy by undergoing experimentally induced cold-pressor test (measured in seconds). Cold pain threshold responses will be compared within-subject in the taper group and between the two groups.
Pain Tolerance Response (in seconds) - Cold Pressor Test | 3 months
  To compare the effects of opioid taper with initiating buprenorphine maintenance therapy by undergoing experimentally induced cold-pressor test (measured in seconds). Cold pain tolerance responses will be compared within-subject in the taper group and between the two groups.
Pain Threshold Response (in seconds) - Quantitative Sensory Test | 3 months
  To compare the effects of opioid taper with initiating buprenorphine maintenance therapy by undergoing experimentally induced quantitative sensory test pain (measured in seconds). Heat pain threshold responses will be compared within-subject in the taper group and between the two groups.
Pain Tolerance Response (in seconds) - Quantitative Sensory Test | 3 months
  To compare the effects of opioid taper with initiating buprenorphine maintenance therapy by undergoing experimentally induced quantitative sensory test pain (measured in seconds). Heat pain tolerance responses will be compared within-subject in the taper group and between the two groups.

SECONDARY OUTCOMES:
Improvement in opioid taper | 3 months
  A sub-aim of the project is to study how the degree of improvement related to opioid taper in experimental pain responses is related to socio-demographic, psychological, and opioid use history characteristic of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Compton, RN, PhD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Avery Road Treatment Center, Rockville, Maryland
  - Kolmac Clinic, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johannes CB, Le TK, Zhou X, Johnston JA, Dworkin RH. The prevalence of chronic pain in United States adults: results of an Internet-based survey. J Pain. 2010 Nov;11(11):1230-9. doi: 10.1016/j.jpain.2010.07.002. Epub 2010 Aug 25. PMID 20797916
- [Background] Chou R, Deyo R, Devine B, Hansen R, Sullivan S, Jarvik JG, Blazina I, Dana T, Bougatsos C, Turner J. The Effectiveness and Risks of Long-Term Opioid Treatment of Chronic Pain. Evid Rep Technol Assess (Full Rep). 2014 Sep;(218):1-219. doi: 10.23970/AHRQEPCERTA218. PMID 30313000
- [Background] Von Korff MR. Long-term use of opioids for complex chronic pain. Best Pract Res Clin Rheumatol. 2013 Oct;27(5):663-72. doi: 10.1016/j.berh.2013.09.011. Epub 2013 Oct 5. PMID 24315147
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on Research Standards for Chronic Low Back Pain. Int J Ther Massage Bodywork. 2015 Sep 1;8(3):16-33. doi: 10.3822/ijtmb.v8i3.295. eCollection 2015 Sep. PMID 26388962
- [Background] The Management of Opioid Therapy for Chronic Pain Working Group. (2010). VA/DOD Clinical Practice Guideline for Management of Opioid Therapy for Chronic Pain. Dept of Veterans Affairs, Department of Defense.
- [Background] Nuckols TK, Anderson L, Popescu I, Diamant AL, Doyle B, Di Capua P, Chou R. Opioid prescribing: a systematic review and critical appraisal of guidelines for chronic pain. Ann Intern Med. 2014 Jan 7;160(1):38-47. doi: 10.7326/0003-4819-160-1-201401070-00732. PMID 24217469
- [Background] Executive Office of the President of the United States of America. (2011). Epidemic: Responding to America's Prescription Drug Abuse. Retrieved January 18, 2016, from White House Website: https://www.whitehouse.gov/sites/default/files/ondcp/policy-and-research/rx_abuse_plan.pdf.
- [Background] Silverman SM. Opioid induced hyperalgesia: clinical implications for the pain practitioner. Pain Physician. 2009 May-Jun;12(3):679-84. PMID 19461836
- [Background] Brush DE. Complications of long-term opioid therapy for management of chronic pain: the paradox of opioid-induced hyperalgesia. J Med Toxicol. 2012 Dec;8(4):387-92. doi: 10.1007/s13181-012-0260-0. PMID 22983894
- [Background] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Background] Mao J. Opioid-induced abnormal pain sensitivity: implications in clinical opioid therapy. Pain. 2002 Dec;100(3):213-217. doi: 10.1016/S0304-3959(02)00422-0. No abstract available. PMID 12467992
- [Background] Compton P, Charuvastra VC, Kintaudi K, Ling W. Pain responses in methadone-maintained opioid abusers. J Pain Symptom Manage. 2000 Oct;20(4):237-45. doi: 10.1016/s0885-3924(00)00191-3. PMID 11027904
- [Background] Compton P, Charuvastra VC, Ling W. Pain intolerance in opioid-maintained former opiate addicts: effect of long-acting maintenance agent. Drug Alcohol Depend. 2001 Jul 1;63(2):139-46. doi: 10.1016/s0376-8716(00)00200-3. PMID 11376918
- [Background] Doverty M, White JM, Somogyi AA, Bochner F, Ali R, Ling W. Hyperalgesic responses in methadone maintenance patients. Pain. 2001 Feb 1;90(1-2):91-6. doi: 10.1016/s0304-3959(00)00391-2. PMID 11166974
- [Background] Eyler EC. Chronic and acute pain and pain management for patients in methadone maintenance treatment. Am J Addict. 2013 Jan;22(1):75-83. doi: 10.1111/j.1521-0391.2013.00308.x. PMID 23398230
- [Background] Pud D, Cohen D, Lawental E, Eisenberg E. Opioids and abnormal pain perception: New evidence from a study of chronic opioid addicts and healthy subjects. Drug Alcohol Depend. 2006 May 20;82(3):218-23. doi: 10.1016/j.drugalcdep.2005.09.007. Epub 2005 Oct 17. PMID 16229972